CLINICAL TRIAL: NCT01851096
Title: A Phase 1, Open-label, Dose-escalation Study of SNX 5422 and Erlotinib in Subjects With Lung Adenocarcinoma With "Acquired Resistance" to Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitors.
Brief Title: Safety and Pharmacology Study of SNX-5422 in Subjects With Resistant Lung Adenocarcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Esanex Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNX-5422-CLN1-007
Record Dates: First submitted 2013-05-04; First posted 2013-05-10 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Cancer
Keywords: Hsp90; SNX-5422; Erlotinib; Lung adenocarcinoma
MeSH Terms: conditions — Neoplasms; Adenocarcinoma of Lung | interventions — SNX-5422

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SNX-5422 (Experimental): Open label administration of SNX-5422 tablets every other day for 21 days on a 28 day cycle. Dose escalation of SNX-5422 based on safety outcomes
  Interventions: Drug: SNX-5422

INTERVENTIONS:
Drug: SNX-5422 — Capsules dosed every other day in the morning starting at a dose of 50 mg/m2. Dose escalation based on safety. Subjects will also receive 150 mg erlotinib daily (in the afternoon).

SUMMARY:
Heat shock protein 90 (Hsp90) is a chemical in the body that is involved in the promotion of cancer. SNX-5422 is an experimental drug that blocks Hsp90.

DETAILED DESCRIPTION:
Heat shock protein 90 (Hsp90) chaperone proteins stabilize many client proteins including mutant EGFR, and are also hypothesized to help maintain the malignant phenotype of mutant EGFR in lung adenocarcinoma. Treatment of EGFR mutant cell lines with the Hsp90 inhibitor geldanamycin results in cellular degradation, decreased levels of pAKT/cyclin D1, and increased apoptosis. Furthermore, Hsp90 inhibitors hamper growth of tumors in nude mice with gefitinib-resistant H1975-xenografts in vivo.

Clinical data showed that mono-therapy with some Hsp90 inhibitors provides stable disease and some patients have partial remissions as best responses in heavily pre-treated non small cell lung cancer patients.

SNX-5422 is a pro-drug of SNX-2112, a potent, highly selective, small-molecule inhibitor of the molecular chaperone Hsp90. Inhibitors of the chaperone protein Hsp90 are of current interest because of the central role that Hsp90 plays in the maturation and maintenance of numerous proteins, for example HER2 and mutated EGFR, that are critical for tumor cell viability and growth.

ELIGIBILITY:
Inclusion Criteria:

* Males or non-pregnant, non-breastfeeding females 18 years-of-age or older.
* Received treatment with erlotinib/gefitinib throughout the one month prior to enrollment and at least six months at any time.
* Must have undergone a biopsy after the development of acquired resistance.
* Pathologic evidence of advanced lung adenocarcinoma (stage IIIB or stage IV) confirmed histologically/cytologically
* Radiographic progression by RECIST during treatment with erlotinib/gefitinib.
* Measurable (RECIST) indicator lesion not previously irradiated.
* No more than 4 prior lines of cytotoxic chemotherapy, including erlotinib/gefitinib
* Karnofsky performance score ≥70.
* Adequate baseline laboratory assessments, including

  * Absolute neutrophil count (ANC) ≥1.5 x 109/L.
  * WBC >3000/microliter
  * Platelet count of ≥100 x 109/L.
  * Total bilirubin level ≤1.5 times institutional upper limit of normal (ULN), alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤1.5 x ULN.
  * Hemoglobin ≥9 mg/dL.
  * Creatinine <1.5 X upper limit of normal or estimated plasma creatinine clearance of ≥40 mL/min (using the Cockroft-Gault equation)
* Signed informed consent form (ICF).
* Subjects with reproductive capability must agree to practice adequate contraception methods.
* Adequate venous access.

Exclusion Criteria:

* CNS metastases which are symptomatic and /or requiring escalating doses of steroids.
* Prior treatment with any Hsp90 inhibitor.
* Conventional chemotherapy, radiation or monoclonal antibodies within 4 weeks (erlotinib/gefitinib therapy within the past 4 weeks IS allowed).
* Palliative radiation within 2 weeks.
* The need for treatment with medications with clinically-relevant metabolism by the cytochrome P450 (CYP) 3A4 isoenzyme within 3 hours before or after administration of SNX-5422
* Screening ECG QTc interval ≥470 msec for females, ≥450 msec for males.
* At increased risk for developing prolonged QT interval, including hypokalemia or hypomagnesemia, unless corrected to within normal limits prior to first dose of SNX-5422; congenital long QT syndrome or a history of torsade de pointes; currently receiving anti-arrhythmics or other medications that may be associated with QT prolongation.
* Patients with chronic diarrhea or with grade 2 or greater diarrhea despite maximal medical management.
* Gastrointestinal diseases or conditions that could affect drug absorption, including gastric bypass.
* Gastrointestinal diseases that could alter the assessment of safety, including irritable bowel syndrome, ulcerative colitis, Crohn's disease, or hemorrhagic coloproctitis.
* History of documented adrenal dysfunction not due to malignancy.
* Known seropositive for human immunodeficiency virus (HIV) or hepatitis C virus (HCV).
* History of chronic liver disease.
* Active hepatitis A or B.
* Current alcohol dependence or drug abuse.
* Use of an investigational treatment from 30 days prior to the first dose of SNX-5422 and during the study.
* Glaucoma, retinitis pigmentosa, macular degeneration, or any retinal changes detected by ophthalmological examination.
* Other serious concurrent illness or medical condition.
* Psychological, social, familial, or geographical reasons that would hinder or prevent compliance with the requirements of the protocol or compromise the informed consent process.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-03; Primary Completion 2015-10 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Number of patients with dose limiting toxicities | Day 28 of first dose cycle
  Number of patients with dose limiting toxicities defined as adverse events (AE) or laboratory abnormalities of Common Terminology Criteria for Adverse Events(CTCAE) version 4.03 ≥ Grade 3 that are not clearly related to disease progression

SECONDARY OUTCOMES:
Tumor response | Weeks 4, 12, 20 and 28
  Tumor progression relative to baseline; assessment of tumor response will be performed using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
Changes in vital signs, physical examination or clinical laboratory from baseline | Weeks 4, 8, 12, 16, 20, 24 and 28
  Descriptive summaries of vital signs, physical examination and quantitative clinical laboratory changes will be presented by treatment received and study visit. Laboratory toxicities will be graded by severity using common terminology criteria for adverse events (CTCAE) Version 4.03. Frequency and percentage of subjects experiencing clinically relevant toxicities will be summarized by treatment received. Summaries may be repeated by treatment cycle.
Number of patients with ophthalmological changes from baseline | Weeks 4, 16 and 28
  Ophthalmologic assessments (visual acuity, visual field, ophthalmoscopy, dark adaptation, optical coherence tomography) will be presented by cohort, study visit and dose. Number of subjects experiencing clinically relevant changes from baseline in any of these examinations will be presented using descriptive summary

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: No
Phase 1 pharmacology study